CLINICAL TRIAL: NCT05877508
Title: An Exploratory, Randomized, Double-Blind Placebo-Controlled Study to Assess the Safety of an Anti-SARS-CoV-2 Monoclonal Antibody and Response to Treatment in Individuals With Long COVID (outSMART-LC)
Brief Title: Anti-SARS-CoV-2 Monoclonal Antibodies for Long COVID (COVID-19)
Acronym: outSMART-LC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Michael Peluso, MD (Other)
Collaborators: Aerium Therapeutics (Unknown); Patient-Led Research Collaborative (Unknown); PolyBio Research Foundation (Other)
Responsible Party: Sponsor-Investigator, Michael Peluso, MD, Assistant Professor, Medicine, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23-38629
Record Dates: First submitted 2023-05-24; First posted 2023-05-26 (Actual); Results first posted 2025-10-28 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Long COVID; Post-Acute Sequela of COVID-19; Post-Acute COVID-19
Keywords: COVID-19; Long COVID; Post-acute Sequelae of SARS-CoV-2 infection
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- AER002 (Experimental): AER002 1200mg administered once by IV
  Interventions: Drug: AER002
- Placebo (Placebo Comparator): Placebo administered once by IV
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AER002 — Intravenous infusion of AER002
  Arms: AER002
Other: Placebo — Placebo infusion
  Arms: Placebo

SUMMARY:
Persistent viral infection with viral reservoirs and detection of circulating spike protein after the initial acute illness is one potential pathogenic mechanism for Long COVID. This mechanism may be able to be targeted by SARS-CoV-2 monoclonal antibodies (mAbs). This trial will study the safety and efficacy of AER002 to treat individuals with Long COVID in an adult population.

DETAILED DESCRIPTION:
The study will enroll approximately 30 participants who meet the World Health Organization (WHO) Long COVID criteria, with Long COVID attributed to a SARS-CoV-2 variant susceptible to AER002. Participants will be enrolled at a single center and randomized 2:1 to receive a SARS-CoV-2 monoclonal antibody (AER002) 1200mg or placebo. Evaluations will take place at baseline and at timepoints up to 1-year post-infusion.

ELIGIBILITY:
Key Inclusion Criteria (note, additional eligibility criteria not listed here will be assessed at Screening):

* Male, female, or transgender ≥18 years of age at Screening.
* History of confirmed acute SARS-CoV-2 infection.
* Long COVID attributed to a SARS-CoV-2 infection with a variant against which AER002 is known to have neutralizing activity (prior to August 15, 2022). Note: While individuals re-infected with SARS-CoV-2 after August 15, 2022 will not be excluded, the SARS-CoV-2 infection after which Long COVID symptoms began must pre-date August 15, 2022.
* At least two symptoms that are new or worsened since the time of SARS-CoV-2 infection, not known to be attributable to another cause upon assessment by the PI. Symptoms must have been present for at least 60 days prior to screening and must be reported to be at least somewhat bothersome.
* Body mass index (BMI) 18 to 50 kilograms/meter squared (kg/m2), inclusive, at the time of screening.
* Participants who are of childbearing potential (CBP) and male participants with sexual partner(s) who are females of CBP must agree to use adequate contraception from study consent through 360 days after dosing.

Key Exclusion Criteria (note, additional eligibility criteria not listed here will be assessed at Screening):

* Long COVID attributed to a SARS-CoV-2 infection after August 15, 2022.
* Previously received treatment or prophylaxis with a SARS-CoV-2-specific mAb, or plan to receive such treatment before exiting the study.
* Previously received COVID-19 convalescent plasma treatment within 60 days prior to Day 0 or plan to receive such treatment before exiting the study.
* Plans to receive any investigational or approved vaccine or booster for SARS-CoV-2 within 60 days prior to Day 0 or before Day 30 following Day 0.
* Active cardiovascular disease or recent (within 3 months) stroke.
* Recent (within 6 months) or planned major surgery.
* Currently hospitalized or recent (within 1 month) unplanned hospitalization.
* Active Hepatitis Bor C infection .
* Untreated or unstable HIV infection (two or more consecutive plasma HIV RNA values >48 copies/mL in the 6 months prior to screen).
* Severe coagulopathy (international normalized ratio ((INR) >2.0, history of hemophilia).
* Severe anemia (hemoglobin <9 grams/deciliter (g/dL)).
* Moderate or severe immunocompromise, according to the current NIH COVID-19 Treatment Guidelines as of March 6, 2023.
* History of anaphylaxis or hypersensitivity upon receiving IV antibody infusions, any componenets of the intervention, prescription or non-prescription drugs, or food products in the past.
* Pregnant, breastfeeding, or unwilling to practice birth control abide by the contraception requirements outlined in the inclusion criteria.
* Participation in a clinical trial with receipt of an investigational product within 28 days or 5 half-lives (whichever is longer) prior to Day 0.
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2026-07-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Peluso, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF/Zuckerberg San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peluso MJ, Hanson MR, Deeks SG. Infection-associated chronic conditions: Why Long Covid is our best chance to untangle Osler's web. Sci Transl Med. 2024 Nov 13;16(773):eado2101. doi: 10.1126/scitranslmed.ado2101. Epub 2024 Nov 13. PMID 39536121

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 36 people were randomized and received an infusion.
Period: Overall Study
Arm/Group | AER002 | Placebo
Started | 24 | 12
Completed | 24 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AER002 | Placebo | Total
Number analyzed (Participants) | 24 | 12 | 36
Age, Continuous [Median (Full Range); unit: years] | 42 [22 to 67] | 43 [24 to 72] | 42 [22 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 7 | 20
  Male | 11 | 5 | 16
Days Since Infection To Which Long COVID Symptoms Are Attributed [Median (Full Range); unit: days] | 740 [436 to 1308] | 769 [495 to 1322] | 740 [436 to 1322]
BMI at Baseline [Count of Participants; unit: Participants]
  <18.5 | 1 | 0 | 1
  18.5-24.9 | 14 | 7 | 21
  25.0-29.9 | 4 | 3 | 7
  >=30 | 5 | 2 | 7
Time Since Most Recent SARS-CoV-2 Infection [Median (Full Range); unit: Days] | 509 [120 to 1308] | 504 [112 to 1080] | 504 [112 to 1308]
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 22 | 11 | 33
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS)-29 Physical Health Summary Score
Description: This measure will evaluate whether there is a difference between treatment with AER002 versus placebo in baseline adjusted mean PROMIS-29 Physical Health Summary Score at Day 90 post-infusion. PROMIS-29 is a validated scale assessing physical function, anxiety, depression, fatigue, sleep disturbance, ability to participate in social activities, and pain. Each domain is scored on a 5-point scale (without any difficulty, with a little difficulty, with some difficulty, with much difficulty, unable to do). A T-score is calculated from each individual domain. A T score of 50 represents the mean for US general adult population, and 10 is the standard deviation. A lower T score indicates worse physical health.
Time Frame: Day 90
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | AER002 | Placebo
Number analyzed (Participants) | 24 | 12
score on a scale | 40.9 [38.3 to 43.5] | 45.0 [41.3 to 48.6]

2. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS)-29 Physical Health Summary Score
Description: This measure will evaluate whether there is a difference between treatment with AER002 versus placebo in baseline adjusted mean PROMIS-29 Physical Health Summary Score at Day 30 and Day 180 post-infusion. PROMIS-29 is a validated scale assessing physical function, anxiety, depression, fatigue, sleep disturbance, ability to participate in social activities, and pain. Each domain is scored on a 5-point scale (without any difficulty, with a little difficulty, with some difficulty, with much difficulty, unable to do). A T-score is calculated from each individual domain. A T score of 50 represents the mean for US general adult population, and 10 is the standard deviation. A lower T score indicates worse physical health.
Time Frame: Day 30 and Day 180
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | AER002 | Placebo
Number analyzed (Participants) | 24 | 12
score on a scale
  Day 30 | 40.7 [38.1 to 43.3] | 41.7 [38.0 to 45.4]
  Day 180 | 41.7 [39.1 to 44.3] | 44.4 [40.7 to 48.0]

3. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS)-29 Mental Health Summary Score
Description: This measure will evaluate whether there is a difference between treatment with AER002 versus placebo in baseline adjusted mean PROMIS-29 Mental Health Summary Score at Day 90 post-infusion. PROMIS-29 is a validated scale assessing physical function, anxiety, depression, fatigue, sleep disturbance, ability to participate in social activities, and pain. Each domain is scored on a 5-point scale (without any difficulty, with a little difficulty, with some difficulty, with much difficulty, unable to do). A T-score is calculated from each individual domain. A T score of 50 represents the mean for US general adult population, and 10 is the standard deviation. A lower T score indicates worse mental health.
Time Frame: Day 90
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | AER002 | Placebo
Number analyzed (Participants) | 24 | 12
score on a scale | 40.7 [37.9 to 43.5] | 45.4 [41.4 to 49.4]

4. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS)-29 Mental Health Summary Score
Description: This measure will evaluate whether there is a difference between treatment with AER002 versus placebo in baseline adjusted mean PROMIS-29 Mental Health Summary Score at Day 30 and Day 180 post-infusion. PROMIS-29 is a validated scale assessing physical function, anxiety, depression, fatigue, sleep disturbance, ability to participate in social activities, and pain. Each domain is scored on a 5-point scale (without any difficulty, with a little difficulty, with some difficulty, with much difficulty, unable to do). A T-score is calculated from each individual domain. A T score of 50 represents the mean for US general adult population, and 10 is the standard deviation. A lower T score indicates worse mental health.
Time Frame: Day 30 and Day 180
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | AER002 | Placebo
Number analyzed (Participants) | 24 | 12
score on a scale
  Day 30 | 40.3 [37.5 to 43.1] | 42.7 [38.7 to 46.7]
  Day 180 | 41.3 [38.4 to 44.1] | 43.8 [39.8 to 47.8]

5. Secondary Outcome: Quality of Life (Global Health Score) 100-point Visual-Analogue Scale
Description: This measure will evaluate whether there is a difference between treatment with AER002 versus placebo in the baseline adjusted mean Quality of Life 100-point Visual-Analogue-Scale at Day 90 post-infusion. 0 represents the worst health a person can imagine and 100 represents the best health a person can imagine.
Time Frame: Day 90
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | AER002 | Placebo
Number analyzed (Participants) | 24 | 12
units on a scale | 53.2 [47.3 to 59.0] | 62.6 [54.3 to 70.9]

6. Secondary Outcome: Quality of Life (5-Item EuroQol EQ-5D-5L) Index Value Score
Description: This measure will evaluate whether there is a difference between treatment with AER002 versus placebo in baseline adjusted mean Quality of Life (5-Item EuroQol EQ-5D-5L) Index Value Score at Day 90 post-infusion. 5-Item EuroQol EQ-5D-5L questions assess pain/difficulty in day-to-day activities over the past week. The 5-Item EuroQol EQ-5D-5L produces a score that typically ranges from 0 - 1, with a higher score indicating better quality of life.
Time Frame: Day 90
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | AER002 | Placebo
Number analyzed (Participants) | 24 | 12
score on a scale | 0.51 [0.42 to 0.61] | 0.67 [0.53 to 0.80]

7. Secondary Outcome: Duke Activity Status Index (DASI)
Description: This measure will evaluate whether there is a difference between treatment with AER002 versus placebo in baseline adjusted mean DASI at Day 90 post-infusion. The Duke Activity Status Index is a patient-reported estimate of functional capacity, maximal oxygen consumption (VO2 max) and maximum metabolic equivalent of tasks (METs). The DASI questionnaire produces a score between 0 and 58.2 points, which is linearly correlated with a patient's VO2 max and METs, as measured from cardiopulmonary exercise testing (CPET). It inquires about a person's ability to perform self-care, walk, climb stairs, run, do house and yard work, engage in sexual intercourse, and perform moderate recreational activities. A higher score indicates higher functional capacity.
Time Frame: Day 90
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | AER002 | Placebo
Number analyzed (Participants) | 24 | 12
score on a scale | 35.6 [31.5 to 39.7] | 40.2 [34.3 to 46.1]

8. Secondary Outcome: Composite Autonomic Symptom Score-31 (COMPASS-31)
Description: This measure will evaluate whether there is a difference between treatment with AER002 versus placebo in baseline adjusted mean COMPASS-31 score at Day 90 post-infusion. COMPASS-31 asks 31 questions related to autonomic dysfunction. The answer to each question generates a numeric score for the question, which is then summed at the end of the questionnaire. A total score out of 100 is generated summarizing orthostatic intolerance, vasomotor, secretomotor, gastrointestinal, urinary, pupillomotor, temperature intolerance, and sexual impairment. The total score ranges from 0 to 100 and a higher score indicates more severe autonomic dysfunction.
Time Frame: Day 90
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | AER002 | Placebo
Number analyzed (Participants) | 24 | 12
score on a scale | 18.3 [13.4 to 23.3] | 13.6 [6.6 to 20.6]

9. Secondary Outcome: World Health Organization Disability Assessment Schedule 2.0 (WHO-DAS 2.0)
Description: This measure will evaluate whether there is a difference between treatment with AER002 versus placebo in baseline adjusted mean WHO-DAS 2.0 score at Day 90 post-infusion. The World Health Organization Disability Assessment Schedule 2.0 questionnaire asks about difficulties due to health conditions. Health conditions include diseases or illnesses, other health problems that may be short or long lasting, injuries, mental or emotional problems, and problems with alcohol or drugs. The range is scored from 0-48, with a higher score indicating a higher level of disability.
Time Frame: Day 90
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | AER002 | Placebo
Number analyzed (Participants) | 24 | 12
score on a scale | 16.9 [14.5 to 19.2] | 12.9 [9.6 to 16.2]

10. Secondary Outcome: Patient Global Impression of Change (PGIC) Scale
Description: This measure will evaluate whether there is a difference between treatment with AER002 versus placebo on the Patient Global Impression of Change (PGIC) scale at Day 90 post-infusion. The self-reported PGIC reflects a patient's belief about the efficacy of treatment. We used a modified PGIC scale which has been used to study pain syndromes and has been employed in other Long COVID clinical trials. It is a common data element developed by the National Institutes of Mental Health. The PGIC ranges from 0 (Much better) to 10 (Much Worse). A score of 5 indicates no change.
Time Frame: Day 90
Measure: Count of Participants; unit: Participants
Arm/Group | AER002 | Placebo
Number analyzed (Participants) | 24 | 12
Participants
  0 - Much Better | 1 | 1
  1 | 0 | 2
  2 | 1 | 2
  3 | 5 | 3
  4 | 6 | 2
  5 - No Change | 7 | 1
  6 | 3 | 0
  7 | 0 | 1
  8 | 1 | 0
  9 | 0 | 0
  10 - Much Worse | 0 | 0

11. Secondary Outcome: Everyday Cognition Form (ECog-39)
Description: This measure will evaluate whether there is a difference between treatment with AER002 versus placebo in baseline adjusted mean ECog-39 score at Day 90 post-infusion. The ECog-39 is an instrument that measures the decline in everyday cognitive and functional abilities that map to six cognitive domains, adapted specifically to describe change in abilities since having COVID. A summary ECog-39 score is calculated scored with a range of 1-4, with a higher score indicating greater cognitive impairment.
Time Frame: Day 90
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | AER002 | Placebo
Number analyzed (Participants) | 24 | 12
score on a scale | 2.09 [1.89 to 2.28] | 1.93 [1.65 to 2.20]

12. Secondary Outcome: 6 Minute Walking Test (6MWT)
Description: This measure will evaluate whether there is a difference between treatment with AER002 versus placebo in baseline adjusted mean distance walked on the 6MWT at Day 90 post-infusion. The 6MWT requires an individual to walk at their normal pace for 6 minutes on a marked track (for example, a hallway). Vital signs are assessed, and the total distance covered is the primary outcome of interest.
Time Frame: Day 90
Measure: Mean (95% Confidence Interval); unit: meters
Arm/Group | AER002 | Placebo
Number analyzed (Participants) | 24 | 12
meters | 426 [400 to 452] | 457 [420 to 495]

13. Secondary Outcome: Active Stand Test
Description: The active standing test is a non-invasive tool to assess orthostatic hypotension (OH) and postural orthostatic tachycardia syndrome (POTS). In short, blood pressure and heart rate measurements were obtained after 5 minutes of resting supine and 1, 3, 5, and 10 minutes of continuous standing. Abnormal active standing test results were defined as those with a decline of >20 mmHg in systolic or > 10 mmHg in diastolic blood pressure in at least two consecutive measurements, or those with an increase in heart rate > 30 bpm on two consecutive measurements.
Time Frame: Day 90
Measure: Count of Participants; unit: Participants
Arm/Group | AER002 | Placebo
Number analyzed (Participants) | 24 | 12
Participants
  Abnormal Active Stand Test | 1 | 0
  Normal Active Stand Test | 23 | 12

14. Secondary Outcome: Neurocognition Index (NCI) Standard Score From the CNS-VS
Description: This measure will evaluate whether there is a difference between treatment with AER002 versus placebo in baseline adjusted mean NCI standard score from the CNS-VS at Day 90 post-infusion. The CNS Vital Signs is a a computer-based neurocognitive assessment comprised of seven tests: verbal and visual memory, finger tapping, symbol digit coding, the Stroop Test, a test of shifting attention and the continuous performance test. The battery gives a summary neurocognition index (NCI) score averaging five domain scores (Composite Memory, Psychomotor Speed, Reaction Time, Complex Attention, and Cognitive Flexibility) and representing a global score of neurocognition. NCI scores are normalized scores (mean 100, standard deviation 15) that are age matched relative to other people in a normative sample. A higher score indicates better cognitive function.
Time Frame: Day 90
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | AER002 | Placebo
Number analyzed (Participants) | 24 | 12
score on a scale | 99.4 [96.8 to 102] | 100.8 [97.2 to 104]

15. Secondary Outcome: C-Reactive Protein (CRP)
Description: This measure will evaluate whether there is a difference between treatment with AER002 versus placebo in baseline adjusted mean CRP concentration (mg/L) at Day 90 post-infusion.
Time Frame: Day 90
Measure: Mean (95% Confidence Interval); unit: mg/L
Arm/Group | AER002 | Placebo
Number analyzed (Participants) | 24 | 12
mg/L | 1.52 [1.03 to 2.00] | 1.37 [.68 to 2.06]

16. Secondary Outcome: Erythrocyte Sedimentation Rate (ESR)
Description: This measure will evaluate whether there is a difference between treatment with AER002 versus placebo in baseline adjusted mean ESR at Day 90 post-infusion.
Time Frame: Day 90
Measure: Mean (95% Confidence Interval); unit: mm/hr
Arm/Group | AER002 | Placebo
Number analyzed (Participants) | 24 | 12
mm/hr | 11.5 [8.88 to 14] | 12.3 [8.70 to 16]

17. Secondary Outcome: D-Dimer
Description: This measure will evaluate whether there is a difference between treatment with AER002 versus placebo in baseline adjusted mean D-Dimer at Day 90 post-infusion.
Time Frame: Day 90
Measure: Mean (95% Confidence Interval); unit: mg/L FEU
Arm/Group | AER002 | Placebo
Number analyzed (Participants) | 24 | 12
mg/L FEU | 0.31 [0.29 to 0.33] | 0.33 [0.29 to 0.36]

18. Secondary Outcome: Fibrinogen
Description: This measure will evaluate whether there is a difference between treatment with AER002 versus placebo in baseline adjusted mean fibrinogen concentration (mg/dL) at Day 90 post-infusion.
Time Frame: Day 90
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | AER002 | Placebo
Number analyzed (Participants) | 24 | 12
mg/dL | 315 [298 to 332] | 299 [275 to 323]

ADVERSE EVENTS:
Time Frame: Up to 12 Months
Description: All gradable SAEs/AEs collected on study, regardless of relatedness to study drug
Arm/Group | AER002 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/12
Other Adverse Events (participants affected / at risk) | 21/24 | 12/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AER002 (N=24) | Placebo (N=12)
Rebound COVID-19 (Infections and infestations) | 0 | 1
Small intestinal bacterial overgrowth (Infections and infestations) | 0 | 1
Suspected oral infection (Infections and infestations) | 0 | 1
Decreased fibrinogen (Blood and lymphatic system disorders) | 2 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Muscle pain/aches (Musculoskeletal and connective tissue disorders) | 6 | 0
Pain at infusion site (Musculoskeletal and connective tissue disorders) | 1 | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pelvic congestion syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Gout flare (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator cuff tear (Musculoskeletal and connective tissue disorders) | 0 | 1
Torn meniscus (Musculoskeletal and connective tissue disorders) | 0 | 1
Torn patellar cartilage (Musculoskeletal and connective tissue disorders) | 0 | 1
Torn pulley ligament (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 1
Trouble with balance/feeling unsteady (Nervous system disorders) | 1 | 1
Brain fog (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Head pressure (Nervous system disorders) | 1 | 0
Intractable chronic migraine with aura (Nervous system disorders) | 1 | 0
Lightheadedness (Nervous system disorders) | 1 | 0
Numbness (Nervous system disorders) | 1 | 0
Abnormal brain MRI (Nervous system disorders) | 0 | 1
Burning sensation in feet (Nervous system disorders) | 0 | 1
Tingling (Nervous system disorders) | 0 | 1
Blurry vision (Eye disorders) | 1 | 0
Keratoconjunctivitissicca (Eye disorders) | 0 | 1
Light sensitivity (Eye disorders) | 0 | 1
Superficial thrombophlebitis (Cardiac disorders) | 1 | 0
Hypertension (Cardiac disorders) | 0 | 1
Hypotension (Cardiac disorders) | 0 | 1
Bruise (Skin and subcutaneous tissue disorders) | 2 | 1
Localized rash (Skin and subcutaneous tissue disorders) | 1 | 0
Skin pain (Skin and subcutaneous tissue disorders) | 1 | 0
Localized itchiness (Skin and subcutaneous tissue disorders) | 0 | 1
Cold sores (Skin and subcutaneous tissue disorders) | 1 | 2
Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic rhinosinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Gastroenteritis (Gastrointestinal disorders) | 2 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 3
Constipation (Gastrointestinal disorders) | 0 | 1
Post-exertional malaise (General disorders) | 3 | 4
Fatigue (General disorders) | 3 | 0
Pre-syncope (General disorders) | 2 | 1
Chills (General disorders) | 1 | 0
Subjective fever (General disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Kidney stone (Renal and urinary disorders) | 1 | 0
Urinary tract infection (Renal and urinary disorders) | 1 | 0
Flank pain (Renal and urinary disorders) | 0 | 1
Non-specific viral infection (Infections and infestations) | 7 | 1
SARS-CoV-2 infection - confirmed (Infections and infestations) | 6 | 4
SARS-CoV-2 infection - suspected (Infections and infestations) | 1 | 2
Skin/soft tissue infection (Infections and infestations) | 1 | 1

LIMITATIONS AND CAVEATS:
This is a small proof-of-concept study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-16): https://cdn.clinicaltrials.gov/large-docs/08/NCT05877508/Prot_SAP_000.pdf